CLINICAL TRIAL: NCT02168816
Title: Efficacy of Oral Antibiotic Therapy Compared to Intravenous Antibiotic Therapy for the Treatment of Diabetic Foot Osteomyelitis (CRO-OSTEOMYELITIS)
Brief Title: Efficacy of Oral Antibiotic Therapy Compared to Intravenous Antibiotic Therapy for Osteomyelitis
Acronym: CRO-OSTEO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was stopped for feasibility (i.e., low recruitment)
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Michael Pinzur, M.D., Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 206209
Record Dates: First submitted 2014-06-10; First posted 2014-06-20 (Estimated); Results first posted 2018-06-08 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: Osteomyelitis
Keywords: Osteomyelitis; Diabetes; Foot Infection
MeSH Terms: conditions — Osteomyelitis; Diabetes Mellitus | interventions — Piperacillin; Tazobactam; Piperacillin, Tazobactam Drug Combination; Cefepime; Metronidazole; Aztreonam; Vancomycin; Daptomycin; Linezolid; Meropenem; Anti-Bacterial Agents; Sulfamethoxazole; Trimethoprim; Trimethoprim, Sulfamethoxazole Drug Combination; Clindamycin; clindamycin phosphate; Moxifloxacin; Ciprofloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Midfoot (Active Comparator): Individuals with an infection on the midfoot are randomized to an intravenous antibacterial agent or an oral antibacterial agent.
  Interventions: Drug: Intravenous Antibacterial Agent; Drug: Oral Antibacterial Agent
- Hindfoot (Active Comparator): Individuals with an infection on the hindfoot are randomized to an intravenous antibacterial agent or an oral antibacterial agent.
  Interventions: Drug: Intravenous Antibacterial Agent; Drug: Oral Antibacterial Agent
- Toe (Active Comparator): Individuals with an infection on the toe are randomized to an intravenous antibacterial agent or an oral antibacterial agent.
  Interventions: Drug: Intravenous Antibacterial Agent; Drug: Oral Antibacterial Agent

INTERVENTIONS:
Drug: Intravenous Antibacterial Agent — Individuals in this arm receive an intravenous antibacterial agent. They are not assigned to specific medications. Individuals in this arm will receive an intravenous antibacterial agent as determined by their primary healthcare provider. This therapy is usually one of the following intravenous medications: (i) piperacillin/tazobactam (Zosyn), (ii) cefepime, (iii) metronidazole, (iv) aztreonam, (v) vancomycin, (vi) daptomycin, (vii) linezolid (Zyvox), and/or (viii) meropenem.
  Other Names: Piperacillin/tazobactam (Zosyn); Cefepime; Metronidazole; Aztreonam; Vancomycin; Daptomycin; Linezolid (Zyvox); Meropenem
Drug: Oral Antibacterial Agent — Individuals in this arm receive an oral antibacterial agent. They are not assigned to specific medications. Individuals in this arm will receive an oral antibacterial agent as determined by their primary healthcare provider. This therapy is usually one of the following oral medications: (i) sulfamethoxazole/trimethoprim (SMX-TMP), (ii) clindamycin (Clindesse), (iii) linezolid (Zyvox), (iv) moxifloxacin (Avelox), (v) ciprofloxacin (Cetraxal), and/or (vi) metronidazole (Flagyl)
  Other Names: Sulfamethoxazole/Trimethoprim (SMX-TMP); Clindamycin (Clindesse); Linezolid (Zyvox); Moxifloxacin (Avelox); Ciprofloxacin (Cetraxal); Metronidazole (Flagyl)

SUMMARY:
The Infectious Diseases Society of America (IDSA) 2012 guidelines for the diagnosis and treatment of diabetic foot infections state that for the treatment of diabetic foot osteomyelitis "No data support the superiority of any specific antibiotic agent or treatment strategy, route, or duration of therapy." Traditionally, osteomyelitis has been treated with a long course of intravenous antibiotics, generally six weeks. Oral antibiotics with high bioavailability and adequate bone penetration have been shown in published studies to be effective for the treatment of osteomyelitis.

The investigators propose to conduct a prospective, single-center, randomized, open trial at Loyola University Medical Center (LUMC) comparing the efficacy of oral antibiotic therapy to intravenous (IV) antibiotic therapy for the treatment of diabetic foot osteomyelitis. The investigators hypothesize that oral antibiotic therapy is equivalent to IV antibiotic therapy. Bone/tissue cultures are obtained for all patients for clinical purposes and are sent to pathology for histologic examination and to the clinical microbiology laboratory for culture and susceptibility. Patients will receive six weeks of IV or oral antibiotic therapy depending upon their randomization group. Primary outcomes at six months clinical follow-up will include: (i) no evidence of bone infection and (ii) resolution of ulcer.

DETAILED DESCRIPTION:
Currently, available literature is not adequate to determine the best agent, route, or duration of antibiotic therapy for the treatment of chronic osteomyelitis. The standard of therapy has been to treat patients with a parenteral antibiotic for four to six weeks. In a recent literature review by Spellberg et al. it was concluded that oral and parenteral antibiotic therapy have similar cure rates for the treatment of chronic osteomyelitis. Oral antibiotic therapy is associated with a lower risk to the patient due to avoiding the need of a central IV line. Additionally, oral therapy costs less than a course of IV antibiotics. Oral antibiotics with high bioavailability and good bone penetration include, fluoroquinolones, linezolid, trimethoprim/sulfamethoxazole (2 tabs bid), clindamycin and metronidazole. These antibiotics have been shown in recent studies to obtain levels in the bone that exceed the minimum inhibitory concentration (MIC) levels of the targeted organisms. According to the IDSA 2012 guidelines for the treatment of diabetic foot infections, the diagnosis of osteomyelitis can be made via plain radiographs or MRI imaging (more sensitive). A bone scan can be considered if an MRI cannot be done. The preferred method of diagnosis is by bone culture and histology. The guidelines also recommend surgical debridement to healthy tissue for diabetic foot infections followed by antibiotic therapy.

The Purpose of this study is to compare the efficacy of oral antibiotic therapy with intravenous antibiotic therapy for the treatment of diabetic foot osteomyelitis following surgical debridement. They hypothesis is that oral antibiotic therapy is equivalent to intravenous antibiotic therapy for the treatment of diabetic foot osteomyelitis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Diagnosis of Diabetes Mellitus (per past medical history documented in the patient medical record)
* Foot osteomyelitis (distal to ankle)
* Surgical debridement (in operating room)

Exclusion Criteria:

* Absolute neutrophil count (ANC) < 500
* Pregnant or lactating patients
* Patients with organisms resistant to oral therapy
* Internal hardware
* Definitive amputations (BKA)
* Limb ischemia [absent pedal pulses or ankle-brachial index (ABI) < 0.5]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03-19 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pinzur, M.D., Principal Investigator — Loyola University
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data

REFERENCES:
- [Background] Lipsky BA, Berendt AR, Cornia PB, Pile JC, Peters EJ, Armstrong DG, Deery HG, Embil JM, Joseph WS, Karchmer AW, Pinzur MS, Senneville E; Infectious Diseases Society of America. 2012 Infectious Diseases Society of America clinical practice guideline for the diagnosis and treatment of diabetic foot infections. Clin Infect Dis. 2012 Jun;54(12):e132-73. doi: 10.1093/cid/cis346. PMID 22619242
- [Background] Spellberg B, Lipsky BA. Systemic antibiotic therapy for chronic osteomyelitis in adults. Clin Infect Dis. 2012 Feb 1;54(3):393-407. doi: 10.1093/cid/cir842. Epub 2011 Dec 12. PMID 22157324
- [Background] Lazzarini L, Lipsky BA, Mader JT. Antibiotic treatment of osteomyelitis: what have we learned from 30 years of clinical trials? Int J Infect Dis. 2005 May;9(3):127-38. doi: 10.1016/j.ijid.2004.09.009. PMID 15840453
- [Background] Bouazza N, Pestre V, Jullien V, Curis E, Urien S, Salmon D, Treluyer JM. Population pharmacokinetics of clindamycin orally and intravenously administered in patients with osteomyelitis. Br J Clin Pharmacol. 2012 Dec;74(6):971-7. doi: 10.1111/j.1365-2125.2012.04292.x. PMID 22486719
- [Background] Wukich DK, Armstrong DG, Attinger CE, Boulton AJ, Burns PR, Frykberg RG, Hellman R, Kim PJ, Lipsky BA, Pile JC, Pinzur MS, Siminerio L. Inpatient management of diabetic foot disorders: a clinical guide. Diabetes Care. 2013 Sep;36(9):2862-71. doi: 10.2337/dc12-2712. PMID 23970716
- [Background] Pinzur MS, Gil J, Belmares J. Treatment of osteomyelitis in charcot foot with single-stage resection of infection, correction of deformity, and maintenance with ring fixation. Foot Ankle Int. 2012 Dec;33(12):1069-74. doi: 10.3113/FAI.2012.1069. PMID 23199855

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from March 2014 through February 2017 (36 months) from a tertiary care practice
Pre-assignment Details: Prior to randomization, 16 participants were excluded because they tested positive for organisms that were resistant to oral antibiotic therapy. Additionally, one participant withdrew prior to randomization and one participant was excluded prior to randomization due to a definitive amputation.
Groups:
- Oral Antibacterial Agent: Individuals in this arm were randomized to an oral antibacterial agent. They were not assigned to specific medications. Instead, individuals in this arm received an oral antibacterial agent as determined by their primary healthcare provider. This therapy was usually one of the following oral medications: (i) sulfamethoxazole/trimethoprim (SMX-TMP), (ii) clindamycin (Clindesse), (iii) linezolid (Zyvox), (iv) moxifloxacin (Avelox), (v) ciprofloxacin (Cetraxal), and/or (vi) metronidazole (Flagyl)
- Intravenous Antibacterial Agent: Individuals in this arm were randomized to an intravenous antibacterial agent. They were not assigned to specific medications. Instead, individuals in this arm received an intravenous antibacterial agent as determined by their primary healthcare provider. This therapy was usually one of the following intravenous medications: (i) piperacillin/tazobactam (Zosyn), (ii) cefepime, (iii) metronidazole, (iv) aztreonam, (v) vancomycin, (vi) daptomycin, (vii) linezolid (Zyvox), and/or (viii) meropenem.
Period: Overall Study
Arm/Group | Oral Antibacterial Agent | Intravenous Antibacterial Agent
Started | 5 | 7
Completed | 3 | 5
Not Completed | 2 | 2
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intravenous Antibacterial Agent | Oral Antibacterial Agent | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 56.18 [36.28 to 70.59] | 45.86 [37.99 to 62.00] | 54.60 [37.14 to 65.03]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 5 | 4 | 9
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 4 | 3 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 12
Comorbid Diabetes [Count of Participants; unit: Participants]
  No | 0 | 0 | 0
  Yes | 7 | 5 | 12
Comorbid Peripheral Vascular Disease [Count of Participants; unit: Participants]
  No | 6 | 5 | 11
  Yes | 1 | 0 | 1
Comorbid Coronary Artery Disease [Count of Participants; unit: Participants]
  No | 6 | 4 | 10
  Yes | 1 | 1 | 2
Comorbid Chronic Kidney Disease [Count of Participants; unit: Participants]
  No | 7 | 4 | 11
  Yes | 0 | 1 | 1
Comorbid Hypertension [Count of Participants; unit: Participants]
  No | 2 | 2 | 4
  Yes | 5 | 3 | 8
Comorbid Heart Disease [Count of Participants; unit: Participants]
  No | 7 | 4 | 11
  Yes | 0 | 1 | 1
Comorbid Hyperlipidemia [Count of Participants; unit: Participants]
  No | 3 | 3 | 6
  Yes | 4 | 2 | 6
Comorbid Thyroid Disorder [Count of Participants; unit: Participants]
  No | 7 | 5 | 12
  Yes | 0 | 0 | 0
Comorbid Depression [Count of Participants; unit: Participants]
  No | 7 | 5 | 12
  Yes | 0 | 0 | 0
Comorbid Cancer [Count of Participants; unit: Participants]
  No | 7 | 5 | 12
  Yes | 0 | 0 | 0
History of Stroke [Count of Participants; unit: Participants]
  No | 7 | 5 | 12
  Yes | 0 | 0 | 0
History of Heart Attack [Count of Participants; unit: Participants]
  No | 7 | 5 | 12
  Yes | 0 | 0 | 0
Comorbid Obesity [Count of Participants; unit: Participants]
  No | 6 | 5 | 11
  Yes | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Bone Infection
Description: Six months following completion of treatment, the researchers record evidence of bone infection for each participant. A negative diagnosis is made when there is (i) an absence of infection based on clinical examination and (ii) down-trending of inflammatory markers. Otherwise, a positive diagnosis is made.
Time Frame: Six Months
Population: The analysis population comprises all randomized participants who had a six month follow-up appointment.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Antibacterial Agent | Oral Antibacterial Agent
Number analyzed (Participants) | 5 | 3
Participants
  Bone Infection Negative | 5 | 3
  Bone Infection Positive | 0 | 0

2. Secondary Outcome: Number of Participants With Ulcer Resolution
Description: Six months following completion of treatment, the researchers record whether each participant's ulcer has resolved.
Time Frame: Six Months
Population: The analysis population comprises all randomized participants who had a six month follow-up appointment.
Measure: Count of Participants; unit: Participants
Arm/Group | Intravenous Antibacterial Agent | Oral Antibacterial Agent
Number analyzed (Participants) | 5 | 3
Participants
  Not Resolved | 5 | 2
  Resolved | 0 | 1

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from March 2014 through February 2017 (36 months)
Arm/Group | Intravenous Antibacterial Agent | Oral Antibacterial Agent
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intravenous Antibacterial Agent (N=7) | Oral Antibacterial Agent (N=5)
Hyperkalemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The trial was stopped prematurely for feasibility (i.e., low recruitment)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT02168816/Prot_SAP_000.pdf